CLINICAL TRIAL: NCT06237036
Title: Clinical Validation of a Computer-Aided Diagnosis (CAD) System Utilizing Artificial Intelligence Algorithms for Continuous and Remote Monitoring of Patient Condition Severity in an Objective and Stable Manner.
Brief Title: Clinical Validation of AI-Based System for Continuous Remote Monitoring of Patient Severity
Acronym: COVIDX_EVCDAO
Status: Completed | Type: Observational
Sponsor: AI Labs Group S.L (Industry)
Collaborators: University Hospital of Torrejon (Other)
Responsible Party: Sponsor
Other Study IDs: LEGIT_COVIDX_EVCDAO_2022
Record Dates: First submitted 2024-01-25; First posted 2024-02-01 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Skin Diseases; Skin Condition
Keywords: Dermatology; Skin lesions; Dermatologist; Artificial Intelligence; Chronic illness
MeSH Terms: conditions — Skin Diseases; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients diagnosed with any of the specified chronic dermatological conditions: The study encompasses patients diagnosed with any of the specified chronic dermatological conditions that meet the inclusion criteria. These patients are attended at the Dermatology Department of the Hospital Universitario de Torrejón.
  Treatment Patients participating in this study did not receive any specific treatment as part of the research protocol.
  Concomitant Medication/Treatment Patients continued their regular prescribed medications and treatments as directed by their primary healthcare providers. No additional medications or treatments were administered as part of this study.
  Follow-Up Duration The follow-up period extended for seven months. Throughout this duration, patients underwent a minimum of two follow-up visits, which could be conducted either remotely or in-person, as per the study's protocol.

SUMMARY:
The goal of this observational prospective and analytical study is to evaluate the effectiveness of the device developed by Legit.Health in remotely monitoring the severity of chronic dermatologic pathologies. Secondly, to assess patient satisfaction with the device for remote monitoring. All this in patients diagnosed with any of the specified chronic dermatological conditions that meet the inclusion criteria. These patients are attended at the Dermatology Department of the Hospital Universitario de Torrejón.

The study proceeded as follows:

Patient Selection and Recruitment Visit The recruitment period spanned six months, during which investigators identified eligible patients. The Principal Investigator (PI) or designated collaborating investigators explained the study details to potential participants using the Patient Information Sheet. Patients had the opportunity to seek clarification on any aspects of the study. If a patient chose to participate, they provided informed consent and received a study code. Data collection commenced post-consent. During this initial visit, patients used the device under the supervision of the research team to complete questionnaires and capture photographs associated with their pathology.

Subsequently, the patient autonomously and remotely continued the data collection process at home, as detailed in the following section.

The device was provided at no cost to patients and the research team for the study's duration.

Procedures Performed by the Patient at Home Completion of Questionnaires Patients independently reported on their condition from home, following instructions provided by the research team and the "Patient Information Guide" integrated into Legit.Health, in conjunction with photograph submissions.

Every two months, patients completed the "Patient Satisfaction Questionnaire" addressing general user experience aspects. Additionally, they completed the System Usability Scale (SUS) Questionnaire at the same frequency

Image capture

Patients simultaneously took photographs of the affected areas while completing questionnaires through the app. These photographs were captured using the patient's smartphone from their homes in an autonomous manner. The frequency of photograph submission was determined by the consulting specialist. No specialized camera equipment was required; patients used the camera available on their smartphones. Patients then transmitted these photographs to the research team through a web app Both patients and members of the medical team possessed access credentials.

The manufacturer did not have access to patient accounts or information. Data transfer and photograph storage adhered to the European Regulation 2016/679 of 27 April on the protection of natural persons with regard to the processing of personal data and the free movement of such data, as well as the Organic Law 3/2018 of 5 December on the Protection of Personal Data and guarantee of digital rights.

DETAILED DESCRIPTION:
Introduction This clinical investigation marks a pivotal stage in the development of the Legit.Health software medical device, designed to enhance dermatological diagnostics using advanced machine vision and deep learning. The study focuses on evaluating the device's effectiveness in remotely monitoring chronic dermatologic conditions and assessing patient satisfaction. With a diverse cohort of 160 patients, rigorous ethical standards, and adherence to regulatory guidelines, this research holds significant potential in revolutionizing dermatological diagnostics.

Objectives Primary objective The primary aim of this study is to ascertain the validity of the device, leveraging artificial intelligence and developed by AI Labs Group S.L., in objectively and reliably tracking the progression of chronic dermatological conditions. This validation is deemed successful if the tool achieves a score of 8 or higher in the Clinical Utility Questionnaire (CUS).

Secondary objectives

In addition to the primary objective, secondary objectives encompass:

Confirming that the utilization of the device elicits a high level of patient satisfaction, particularly in its remote application.

Demonstrating that the implementation of the device leads to a reduction in face-to-face consultations, thereby optimizing healthcare resources and patient convenience.

Validating the device's ability to consistently generate reliable condition monitoring, thereby establishing its trustworthiness as a monitoring system.

Population The study encompasses patients diagnosed with any of the specified chronic dermatological conditions that meet the inclusion criteria. These patients are attended at the Dermatology Department of the Hospital Universitario de Torrejón.

Design and Methods Design

The study proceeded as follows:

1. Patient Selection and Recruitment Visit The recruitment period spanned six months, during which investigators identified eligible patients.

   The Principal Investigator (PI) or designated collaborating investigators explained the study details to potential participants using the Patient Information Sheet. Patients had the opportunity to seek clarification on any aspects of the study.

   If a patient chose to participate, they provided informed consent and received a study code. Data collection commenced post-consent. During this initial visit, patients used the device under the supervision of the research team to complete questionnaires and capture photographs associated with their pathology.

   Subsequently, the patient autonomously and remotely continued the data collection process at home, as detailed in the following section.

   The device was provided at no cost to patients and the research team for the study's duration.
2. Procedures Performed by the Patient at Home 2.1. Completion of Questionnaires Patients independently reported on their condition from home, following instructions provided by the research team and the "Patient Information Guide" (Appendix IV of the protocol) distributed during the screening visit.

At regular intervals, patients documented the status of their pathology using questionnaires and the Dermatology Life Quality Index (DLQI) (Appendix V of the protocol), integrated into Legit.Health, in conjunction with photograph submissions.

Every two months, patients completed the "Patient Satisfaction Questionnaire" (Appendix II of the protocol), addressing general user experience aspects. Additionally, they completed the System Usability Scale (SUS) Questionnaire (Appendix III of the protocol) at the same frequency.

2.2. Image Capture Patients simultaneously took photographs of the affected areas while completing questionnaires through the app. These photographs were captured using the patient's smartphone from their homes in an autonomous manner. The frequency of photograph submission was determined by the consulting specialist. No specialized camera equipment was required; patients used the camera available on their smartphones.

Patients then transmitted these photographs to the research team through a web app (Appendix VII of the protocol). Both patients and members of the medical team possessed access credentials.

The manufacturer did not have access to patient accounts or information. Data transfer and photograph storage adhered to the European Regulation 2016/679 of 27 April on the protection of natural persons with regard to the processing of personal data and the free movement of such data, as well as the Organic Law 3/2018 of 5 December on the Protection of Personal Data and guarantee of digital rights.

Number of Subjects A total of 160 patients were recruited in this study.

Initiation Date March 03rd, 2022

Completion Date October 23rd, 2023

Duration The study spanned a total duration of 19 months, encompassing the time needed for tasks such as database closure and editing, data analysis, and the preparation of the final study report after the recruitment of the last subject.

Methods The study employed a prospective observational analytical design to evaluate the effectiveness of the device in remotely monitoring chronic dermatologic pathologies. The research encompassed a diverse cohort of 160 patients with various dermatological conditions. Data collection involved questionnaires, photograph analysis, and patient satisfaction surveys. The study adhered to strict ethical guidelines, ensuring patient confidentiality and compliance with international standards. Patients were provided with detailed information and informed consent. The study's robust methodology aimed to assess the clinical utility and usability of the device.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided their informed consent for participation in the study.
* Patients who demonstrate proficiency in both written and spoken Spanish or English.
* Patients who possess a smartphone, defined as a phone equipped with internet access and an integrated camera, regardless of make, model, or technical specifications.

Exclusion Criteria:

* Patients who, as determined by the investigator, did not adhere to the study procedures.
* Patients who were already utilizing the tool under investigation prior to the commencement of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with any of the specified chronic dermatological conditions that meet the inclusion criteria. These patients are attended at the Dermatology Department of the Hospital Universitario de Torrejón. It encompassed a diverse patient cohort with a range of chronic dermatologic pathologies, providing a comprehensive representation of the population affected by these conditions.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Malignancy | through study completion, an average of 1 year
  Malignancy of the lesion detected by the tool
Utility | At the end of the study, up to 1 month
  Utility of the application referred by the clinicians

SECONDARY OUTCOMES:
Sex and age | through study completion, an average of 1 year
  Sex and age of patients
Diagnosis | through study completion, an average of 1 year
  Clinical data: diagnosis, date of diagnosis, medication the patient is taking.
Quality of life noticed by patients | through study completion, an average of 1 year
  Quality of life: score of the Dermatology Life Quality Index (DLQI). The questionnaire consists of 10 questions with four alternative answers: "not at all", "a little", "a lot", or "very much" with corresponding scores of 0, 1, 2, and 3, respectively. The response "not relevant" is scored as "0". The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the greater the impairment in quality of life. The DLQI can also be expressed as a percentage of the maximum possible score of 30.
Satisfaction of patients | At the time of recruitment of the last patient in the study, up to 4 weeks
  Degree of patient satisfaction using the patient satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marta Andreu, MD, Principal Investigator — Torrejón University Hospital
Locations (1):
- Torrejón University Hospital, Torrejón de Ardoz, Madrid, Spain